CLINICAL TRIAL: NCT02002377
Title: The SHIFT-2 Study: Use of Intravitreal Aflibercept in Wet Age Related Macular Degeneration (AMD) Patients With an Incomplete Response to Routine Ranibizumab Injections
Brief Title: Intravitreal Aflibercept in Wet Age Related Macular Degeneration Patients With an Incomplete Response to Routine Ranibizumab Injections
Acronym: SHIFT-2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate enrollment due to investigational product becoming newly available on the Canadian market soon after study start
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Age Related Macular Degeneration
Keywords: Age Related Macular Degeneration, wet; aflibercept
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Experimental): Aflibercept 2 mg (0.05 mL or 50 microliters) will be administered by intravitreal injection every 4 weeks for the first 8 weeks, followed by 2 mg (0.05 mL) via intravitreal injection once every 8 weeks for 36 weeks
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Aflibercept 2 mg (0.05 mL or 50 microliters) will be administered by intravitreal injection every 4 weeks for the first 8 weeks, followed by 2 mg (0.05 mL) via intravitreal injection once every 8 weeks for 36 weeks

SUMMARY:
SHIFT-2 is a national, multi-center, non-randomized, open label trial of aflibercept in patients with wet age related macular degeneration who have incomplete response with routineranibizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

Note: Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study

1. Age >50 years
2. Active primary subfoveal choroidal neovascularization (CNV) lesions secondary to AMD including juxtafoveal lesions that affect the fovea as evidenced by Fluorescein Angiography in the study eye
3. Presence of intra or sub retinal fluid on SDOCT in the study eye
4. Current treatment with uninterrupted routine (q35 +/- 7 days) ranibizumab started at least 3 months before Baseline (Week 0), having received at least 3 consecutive ranibizumab injections and no more than 24 injections maximum, with all ranibizumab injection intervals being 35 +/- 7 days apart
5. ETDRS BCVA 20/30 and 20/320 (letter score of 78 to 25) in the study eye

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Presence of purely serous pigment epithelial detachment in the study eye
2. Any scarring or fibrosis involving the center of the fovea in the study eye
3. Prior ocular or systemic treatment/surgery for wet AMD other than ranibizumab IVI monthly (in study the eye)
4. Prior prn or treat and extend treatment with ranibizumab IVI between 3 to 24 months before Baseline (Week 0) in the study eye
5. Prior treatment with systemic anti-VEGF therapy within the last 6 months in the study eye
6. History of vitreous hemorrhage within the last 6 months in the study eye
7. Prior vitrectomy in the study eye
8. History of retinal detachment in the study eye
9. History of macular hole of stage 2 and above in the study eye
10. Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
11. Any intraocular or periocular surgery/invasive procedure during the previous 6 months except lid surgery in the study eye
12. Prior trabeculectomy or other filtration surgery in the study eye
13. Uncontrolled glaucoma (≥ 25mmHg despite treatment with anti-glaucoma medications) in the study eye
14. Aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of a yttrium aluminum garnet (YAG) posterior capsulotomy) in the study eye.
15. Scheduled for intraocular surgery during the study period in the study eye
16. Concurrent retinal disease (i.e. diabetic retinopathy, retinal vein occlusion, retinal detachment, uveitis) in the study eye
17. History of ocular or periocular infection/inflammation in the study eye within the last 4 weeks of screening
18. Pregnant or breastfeeding

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
'OCT defined success' defined by no presence of intra or sub retinal fluid on SDOCT | After 12 weeks of treatment

SECONDARY OUTCOMES:
'OCT defined success' defined by no presence of intra or sub retinal fluid on SDOCT | 16 weeks after treatment
Change in central retinal thickness (CRT) | Weeks 12, 16, and 48
Change in Early Treatment Diabetic Retinopathy Study best-corrected visual acuity | Week 12, 16, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Brent, MD, FRCSC, Principal Investigator — Unity Health Toronto; Rajeev Muni, MD, FRCSC, Principal Investigator — Unity Health Toronto
Locations (9):
- Canada (9):
  - Calgary Retina Consultants, Calgary, Alberta
  - Alberta Retina Consultants, Edmonton, Alberta
  - Capital District Health Authority, Halifax, Nova Scotia
  - St. Joseph's Centre for Ambulatory Services, Hamilton, Ontario
  - Hotel Dieu Hospital / Queen's, Kingston, Ontario
  - Ivey Eye Institute, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Saskatoon Retina Consultants, Saskatoon, Saskatchewan